CLINICAL TRIAL: NCT01644279
Title: Claude D. Pepper Older Americans Independence Center (OAIC); Skeletal Muscle Apoptosis and Physical Performance; Oxidative RNA/DNA Damage and Repair in Aged Human Muscle
Brief Title: Skeletal Muscle Apoptosis and Physical Performance; Oxidative RNA/DNA Damage and Repair in Aged Human Muscle
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 429-2005; 2P30AG028740 (NIH)
Record Dates: First submitted 2012-07-05; First posted 2012-07-19 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Sarcopenia
Keywords: aging; sarcopenia; mitochondria; skeletal muscle; apoptosis
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skeletal muscle biopsy; plasma, serum, urine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Young: Young (age 20-35 years old)
- Old high-functioning: Old high-functioning (age 70-99 years old)
- Old low-functioning: Old low-functioning (age 70-99 years old)

SUMMARY:
The age-related loss of muscle mass and strength, also termed sarcopenia, is a commonly recognized consequence of aging and has been associated with frailty, functional loss, hospitalization, and increased mortality among older people. Sarcopenia and its consequences have a considerable economic impact, since it has been estimated that the healthcare cost attributable to sarcopenia in the US in 2000 was $ 18.5 billions. Preclinical animal models strongly suggest that apoptosis, a programmed cell death, might play a prominent role in the age-related muscle wasting. In specific aim one, the investigators will assess the extent of muscle apoptosis in muscle biopsies obtained from the vastus lateralis muscle of young control subjects (ages 20-35) and high-performance and low-performance older subjects (age range 70-99 years). In specific aim 2, the investigators will investigate the role of Poly (ADP-ribose) polymerase 1 (PARP-1) and apoptosis-inducing factor (AIF) in the induction of skeletal muscle apoptosis. In specific aim 3, the investigators propose to investigate the contribution of the muscle energy deficit, due to the age-related mitochondrial dysfunction, in the development of muscle wasting. Finally, in specific aim 4, the investigators propose to reassess after four years physical performance, muscle mass and the extent of muscle apoptosis, in the high-performing participants, in order to correlate eventual decline in physical function, muscle mass and functional status, with changes in muscle apoptosis and in biochemical parameters in this very old population. Physical performance will be established according to the summary performance score obtained in the Short Form Physical Performance Battery (SPPB). In addition to the SPPB the investigators will also employ hand grip strength and knee extensor strength tests and the investigators will quantify muscle contractile area using 3D magnetic resonance imaging. Disability will be assessed using a self-report questionnaire. These studies will enhance our understanding of the biology and pathophysiology underlying the geriatric syndrome of sarcopenia and provide significant and novel insights that will enable us to identify new potential targets for interventions aimed at preventing and treating sarcopenia and functional impairment in older adults.

DETAILED DESCRIPTION:
Specific Aims:

Specific Aim 1. To determine the extent of muscle apoptosis during aging in young healthy controls and in high-functioning and low-functioning older subjects. The investigators hypothesize that the observed level of muscle cell apoptosis is associated with physical disability. The investigators will recruit a cohort of ten young control subjects (age 20-35). The investigators will also recruit and stratify a cohort of forty elderly (age 70-99 years) into two distinct categories by set criteria based on their level of physical performance. Subjects with a summary performance score ≥ 11 at the Short Physical Performance Battery (SPPB) (66) will be considered high-functioning. Conversely, subjects with a summary performance score ≤ 7 will be considered low-functioning. In addition to the SPPB, the investigators will also perform the hand grip strength test and the isokinetic knee extensor test, and will implement 3D magnetic resonance imaging (MRI) to precisely quantify the quadriceps contractile area. The investigators will obtain a muscle biopsy for each subject to determine the severity of apoptosis using biochemical and histological analyses (see Methods). Disability will be assessed using a self-report questionnaire. Hence, the investigators will determine the extent muscle apoptosis and the investigators will be able to correlate this to the level of physical disability and muscle mass.

Specific Aim 2. To elucidate the role of Poly(ADP-ribose) polymerase 1 (PARP-1) and apoptosis-inducing factor (AIF) in the induction of apoptosis in human skeletal muscle. The investigators hypothesize that the observed cell loss due to apoptosis is mainly related to a caspase-independent mechanism. The investigators have recently shown that activation of mitochondrial caspase-independent pathway of apoptosis may play a more important role than the caspase-dependent pathway in contributing to nuclear cell death (67). Furthermore, the investigators hypothesize that the PARP-1/AIF pathway of apoptosis might be involved in the age-related muscle wasting process. The investigators will quantitatively assess PARP-1 and AIF and correlate these measures with the extent of muscle apoptosis.

Specific Aim 3. To assess the role of mitochondria dysfunction and energy failure in muscle apoptosis, sarcopenia, and disability. The investigators hypothesize that mitochondrial dysfunction and the resulting reduced production of adenosine triphosphate (ATP) is causally related to sarcopenia, possibly by triggering the apoptosis program. It has been estimated that the mean ATP production in the quadriceps muscle of old human subjects is approximately 50% of that of younger subjects (68), and it has been postulated that energy failure might trigger apoptosis (58). Consistently with these findings, the investigators have recently found that in rats' gastrocnemius muscle, ATP content and the rate of ATP production declined by ~50% with age (59). The investigators will quantitatively assess myocytes' ATP content along with key mitochondrial metabolic enzymes, namely citrate synthase, cytochrome-c-oxidase (COX), ATPase, and aconitase. The investigators will correlate these parameters with the level of apoptosis and with measures of physical performance, disability, and muscle mass.

Specific Aim 4. To correlate changes in physical function and muscle mass with muscle apoptosis and biochemical parameters at follow-up (longitudinal study). After 4 years subjects in the high-performance group will be reevaluated for muscle apoptosis rate, PARP-1 and AIF activity, and energy production. The investigators will correlate these parameters with measures of physical performance and muscle mass assessed by MRI, as well as with self-reported disability. Hence, the investigators will be able to directly correlate an eventual decline in physical performance, muscle mass and functional status at this very old age with changes in muscle apoptosis and in biochemical parameters.

Research Plan:

Using a cross-sectional design (age 20-35 and 70-99 years) the investigators will quantify the level of apoptosis in the vastus lateralis muscle in a healthy (see inclusion/exclusion criteria) population. Apoptosis of irreplaceable post-mitotic cells may be important mechanism in the development of sarcopenia and has not been investigated in healthy humans with age. A variety of chronic diseases have documented cases of apoptosis in human skeletal muscle; i.e., chronic pulmonary diseases (69,70) and patients with heart failure (69,71,72). However, it is essential to establish baseline levels of apoptosis in relatively healthy humans before proceeding to more complex conditions, such as disease conditions and frailty. In addition, the investigators will determine knee extensors strength, the myocyte volume, extra cellular space and the myonuclear domain (cross-sectional muscle area/nucleus) by quantifying the number of nuclei within a cross-sectional area of muscle. This specific aim will establish baseline levels of apoptosis and assess standard measures to assess sarcopenia.

Study design. To accomplish our aims, the investigators propose two separates, yet complementary studies

1. In order to gain insights into changes of the apoptosis potential with age and its contribution to muscle mass and strength loss, the investigators will quantify the level of apoptosis in the vastus lateralis muscle in young (age 20-35 years; N =20), old high-functioning, (age 70-99 years; N = 25), and old low-functioning (age 70-99 years; N = 20) subjects. Muscle biopsy and MRI scan to quantify quadriceps contractile area will be performed in the study participants. Muscle strength will be assessed by hand grip strength test and the isokinetic knee extensor test.
2. Preliminary data on the contribution of skeletal muscle apoptosis to sarcopenia, physical function loss in advanced age will be gathered by quantifying the extent of muscle apoptosis in the vastus lateralis muscle of old (age 70-99 years), high-functioning (N = 25) and low-functioning (N = 20) subjects, along with measures of muscle mass (MRI), muscle strength (hand grip and knee extension test), and overall physical performance (Short Physical Performance Battery, SPPB (67)). In addition, the investigators will collect preliminary data regarding the role mitochondrial-driven apoptosis in muscle wasting and functional loss at old age.

A brief physical exam will be administered to all study participants, and major biological signs (body weight, standing height, body temperature, blood pressure, and pulse) will be recorded. A basic questionnaire regarding participants' health history will also be administered

After four years the old participants will be reevaluated for physical performance, functional status muscle mass (MRI), muscle apoptosis, and biochemical parameters Disability will also be assessed using a self-report disability questionnaire. In order to gain information regarding changes in physical performance and functional status with time and to maximize retention, an annual visit employing SPPB, hand grip and knee extensor testing, will be scheduled for the old participants.

ELIGIBILITY:
Inclusion criteria. The following inclusion criteria will be adopted to select the study participants:

* males and females aged 20-35 and 70-99 years
* sedentary lifestyle (i.e., the subject has spent less than 20 minutes per week in the past 2 month performing structured physical activity, such as exercising at a gym and/or weight training)
* willing and able to give informed consent.

Exclusion criteria:

* history of smoking in the prior 12 months
* active treatment for cancer or history of cancer in the past 3 years
* congestive heart failure New York Heart Association (NYHA) Class III or IV
* previous stroke with upper and/or lower extremities involvement within the last 6 months
* peripheral vascular disease Fontaine Class III/IV
* History of life-threatening cardiac arrhythmias, stroke, severe Parkinson's disease or severe neurological disorders likely to interfere with physical function
* cognitive impairment (i.e., Mini-Mental State Examination (MMSE) ≤ 23)
* renal disease requiring dialysis
* lung disease requiring steroids
* lower extremity amputation
* severe osteoarthritis that interferes with physical function
* Complicated diabetes
* inflammatory diseases such as active rheumatoid arthritis, vasculitis, autoimmune disorders, and inflammatory bowel disease
* life-threatening illnesses with an estimated life expectancy less than 1 year
* history of drug or alcohol abuse
* taking growth hormone (GH) and/or estrogen replacement therapy
* Testosterone medication
* Anticoagulant therapy
* involved in active weight loss > 5 kg in prior 3 months
* planning to relocate out of the study area in the next 4 years (ages 70-99 only)
* pregnancy
* SPPB score of 8-10
* Lidocaine allergy
* MRI exclusions, such as pregnancy, claustrophobia, heart pacemaker / defibrillator, heart valve prosthesis, aneurysm clip, metallic stent, neurostimulation system, cochlear implants or inner ear prosthesis, insulin pump or other infusion pump, metal slivers in the orbital area/eye socket

Temporary exclusion criteria:

* recent bacterial infection (< 2 weeks)
* acute febrile illness in prior 2 months
* high blood pressure (i.e., BP ≥ 180/110 mm Hg) at the screening visit (subject will be referred to his/her physician and reevaluated after appropriated therapy being instituted)
* major surgery or hip/knee replacement in the past 6 months

Assessment of disability. The uniform measure proposed to use for the assessment of disability will be a self-report disability questionnaire. This questionnaire was developed for the Fitness Arthritis in Seniors Trial (FAST) and since then has been widely used in intervention and observational studies (e.g. ADAPT, REACT-1, OASIS, CHAMP). The questionnaire is not specific to a certain disease and asks about perceived difficulties in general activities of daily living during the last month. Respondents answer for each of the items whether they experience 1) no difficulty, 2) a little difficulty, 3) some difficulty, 4) a lot of difficulty, 5) unable to do or, 6) did not do for other reasons. Answers can be averaged across the items in order to receive an indication of the overall perceived disability burden by a person.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young (age 20-35 years; N =20), old high-functioning, (age 70-99 years; N = 25), and old low-functioning (age 70-99 years; N = 20) subjects.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2006-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Short Form Physical Performance Battery (SPPB) | baseline
  The SPPB is composed by three subtasks: usual gait speed, standing balance and chair stand tests.
Cytochrome c oxidase activity | baseline
  Cytochrome c oxidase (COX) activity measured in permeabilized fibers from muscle biopsy specimens.
Muscle strength | baseline
  Muscle strength will be assessed by hand grip strength test and the isokinetic knee extensor test.
Quadriceps contractile area | baseline
  3D magnetic resonance imaging (MRI) to precisely quantify the quadriceps contractile area
Peroxisome proliferator-activated receptor γ coactivator α (PGC-1α) | baseline
  Major regulator of mitochondrial content and oxidative metabolism in several tissues, including skeletal muscle; measured in muscle biopsy specimens.
Sirtuin 3 (SIRT3) | baseline
  The induction of mitochondrial gene expression and biogenesis is largely controlled by the coordinated actions of various transcriptional and metabolic regulators including Sirtuin 3 (SIRT3); measured in muscle biopsy specimens.
Short Form Physical Performance Battery (SPPB) | 4 years
  The SPPB is composed by three subtasks: usual gait speed, standing balance and chair stand tests.
Cytochrome c oxidase activity | 4 years
  Cytochrome c oxidase (COX) activity measured in permeabilized fibers from muscle biopsy specimens.
Muscle strength | 4 years
  Muscle strength will be assessed by hand grip strength test and the isokinetic knee extensor test.
Quadriceps contractile area | 4 years
  3D magnetic resonance imaging (MRI) to precisely quantify the quadriceps contractile area
Peroxisome proliferator-activated receptor γ coactivator α (PGC-1α) | 4 years
  Major regulator of mitochondrial content and oxidative metabolism in several tissues, including skeletal muscle; measured in muscle biopsy specimens.
Sirtuin 3 (SIRT3) | 4 years
  The induction of mitochondrial gene expression and biogenesis is largely controlled by the coordinated actions of various transcriptional and metabolic regulators including Sirtuin 3 (SIRT3); measured in muscle biopsy specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Leeuwenburgh, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Joseph AM, Adhihetty PJ, Buford TW, Wohlgemuth SE, Lees HA, Nguyen LM, Aranda JM, Sandesara BD, Pahor M, Manini TM, Marzetti E, Leeuwenburgh C. The impact of aging on mitochondrial function and biogenesis pathways in skeletal muscle of sedentary high- and low-functioning elderly individuals. Aging Cell. 2012 Oct;11(5):801-9. doi: 10.1111/j.1474-9726.2012.00844.x. Epub 2012 Jul 9. PMID 22681576
- [Result] Marzetti E, Lees HA, Manini TM, Buford TW, Aranda JM Jr, Calvani R, Capuani G, Marsiske M, Lott DJ, Vandenborne K, Bernabei R, Pahor M, Leeuwenburgh C, Wohlgemuth SE. Skeletal muscle apoptotic signaling predicts thigh muscle volume and gait speed in community-dwelling older persons: an exploratory study. PLoS One. 2012;7(2):e32829. doi: 10.1371/journal.pone.0032829. Epub 2012 Feb 28. PMID 22389725
- [Result] Buford TW, Lott DJ, Marzetti E, Wohlgemuth SE, Vandenborne K, Pahor M, Leeuwenburgh C, Manini TM. Age-related differences in lower extremity tissue compartments and associations with physical function in older adults. Exp Gerontol. 2012 Jan;47(1):38-44. doi: 10.1016/j.exger.2011.10.001. Epub 2011 Oct 12. PMID 22015325
- [Result] Marzetti E, Landi F, Marini F, Cesari M, Buford TW, Manini TM, Onder G, Pahor M, Bernabei R, Leeuwenburgh C, Calvani R. Patterns of circulating inflammatory biomarkers in older persons with varying levels of physical performance: a partial least squares-discriminant analysis approach. Front Med (Lausanne). 2014 Sep 1;1:27. doi: 10.3389/fmed.2014.00027. eCollection 2014. PMID 25593902
- [Result] Wawrzyniak NR, Joseph AM, Levin DG, Gundermann DM, Leeuwenburgh C, Sandesara B, Manini TM, Adhihetty PJ. Idiopathic chronic fatigue in older adults is linked to impaired mitochondrial content and biogenesis signaling in skeletal muscle. Oncotarget. 2016 Aug 16;7(33):52695-52709. doi: 10.18632/oncotarget.10685. PMID 27447862
- See also: University of Florida Claude D. Pepper Older Americans Independence Center (OAIC) — http://aging.ufl.edu/?q=pepper_center